CLINICAL TRIAL: NCT04886349
Title: Platelet-rich Plasma for Thumb Carpometacarpal Joint Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey S. Brault, Principal Investigator, Mayo Clinic
Other Study IDs: 20-008912
Record Dates: First submitted 2021-04-14; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Thumb Carpometacarpal Joint Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Platelet-rich plasma — Platelet-rich plasma injection for first CMC OA

SUMMARY:
The purpose of this study is to investigate a case series of patients treated with Platelet-rich plasma for thumb carpometacarpal joint osteoarthritis. Carpometacarpal arthritis is a highly prevalent condition with significant effects on quality of life and function. Meanwhile, platelet-rich plasma has been demonstrated to be an effective treatment for various musculoskeletal conditions.

DETAILED DESCRIPTION:
The first carpometacarpal (CMC) joint at the base of the thumb is one of the most commonly affected joints by osteoarthritis (OA), with a prevalence ranging from 15-36% in females and 5-11% in males. It is also functionally debilitating, with symptoms including diminished range of motion, weakness, deformity, instability, and pain. Despite the prevalence of first CMC OA, as well as the emerging evidence of platelet-rich plasma (PRP) efficacy for various musculoskeletal conditions, there is a paucity of studies investigating the two. To our knowledge, there are three studies in the literature, resulting in a total of 27 patients with first CMC OA receiving PRP to date1.

Common nonsurgical treatment options for management of this condition include oral and topical NSAIDs, hand therapy, activity modifications, splinting and intra-articular injections. Injections have traditionally consisted of corticosteroids demonstrating variable efficacy and viscosupplementation resulting in conflicting results. Surgical options include trapeziectomy with ligament reconstruction and tendon interposition, fusion, and less commonly, implant arthroplasty.

PRP is defined as an autologous, concentrated mix of platelets and inflammatory mediators suspended in plasma, obtained by centrifuging a patient's whole blood. It is hypothesized that PRP stimulates recruitment, proliferation, and differentiation of regenerative cells via release of various growth factors such as platelet-derived growth factor-AB and -BB, transforming growth factor-β1, insulin-like growth factor-1, fibroblast growth factor-basic, epidermal growth factor, vascular endothelial growth factor, and interleukin (IL)-12. The platelets in PRP have anti-inflammatory properties with modulators including IL-1 receptor antagonist, soluble tumor necrosis factor receptor I and II, IL-4, IL-10, IL-13 and interferon γ. Although PRP has been used for numerous musculoskeletal conditions, varying methods of extraction, different types of PRP, and lack of standardized reporting on the detailed biologic makeup of PRP has caused difficulties with interpretation and comparison of studies investigating its use. For these reasons, there has been a call for the standardization of PRP in clinical use.

The primary aim of this study was to assess (1) outcomes of PRP injection among patients with first CMC OA, and (2) the biologic characteristics of PRP injectate. The secondary aims were to describe the injection technique used at our institution and analyze the relationships between patient demographics, PRP biologic characteristics, and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Patients who previously underwent PRP injection of their first CMC joint.

Exclusion Criteria:

- Individuals less than 18 years of age.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those with CMC OA who received PRP injections
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | up to 12 months
  Subjective patient satisfaction on a 1-5 point scale with 1 being the worst, 5 being the best. Obtained via follow-up interview.
Patient symptom improvement | up to 12 months
  Subjective symptom satisfaction on a 1-5 point scale with 1 being the worst, 5 being the best. Obtained via follow-up interview.
Visual analogue pain scale | up to 12 months
  Subjective pain rating on a scale of 1-10 with 1 being no pain and 10 being severe pain. Obtained via automatically-generated follow-up questionnaire through electronic medical record. Obtained via follow-up interview.
Follow-up procedures/surgeries/interventions | up 12 months
  Patient described any required procedures/surgeries/interventions
Biologic characteristics of the whole blood and platelet-rich plasma included platelets, erythrocytes, leukocytes, neutrophils, lymphocytes, and monocytes | Day of procedure (within 24 hours of procedure)
  Platelets, erythrocytes, leukocytes, neutrophils, lymphocytes, and monocytes were measured in whole blood and platelet-rich plasma. These were reported in concentration of 10^9/milliliter. There is little data regarding these expected values of platelet rich plasma and these are known to vary widely. Obtained through quality control analysis which was sent to pathology lab the day of procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Brault, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials